CLINICAL TRIAL: NCT03196297
Title: A Multi-Centre Trial Evaluating Efficacy and Safety of Prophylactic Administration of Concizumab in Patients With Severe Haemophilia A Without Inhibitors
Brief Title: A Trial Evaluating Efficacy and Safety of Prophylactic Administration of Concizumab in Patients With Severe Haemophilia A Without Inhibitors
Acronym: explorer™5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7415-4255; U1111-1179-3872 (Other: World Health Organization (WHO)); 2016-000614-29 (Registry Identifier: EudraCT); JapicCTI-173682 (Registry Identifier: JAPIC)
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Results first posted 2021-05-10 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Haemostasis; Haemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — concizumab; recombinant factor VIII N8

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Concizumab (Experimental): Daily administration of concizumab to both on-demand and prophylaxis patients
  Interventions: Drug: Concizumab; Drug: Turoctocog alfa

INTERVENTIONS:
Drug: Concizumab — 0.15 mg/kg (with potential stepwise dose administration to 0.25 mg/kg) administered daily s.c (subcutaneously, under the skin). Treatment duration is 24 weeks in the main phase, and 52 weeks in the extension phase
Drug: Turoctocog alfa — Breakthrough bleeding episodes will be treated by the patients at home with turoctocog alfa at the discretion of the study doctor, who will also choose dose levels

SUMMARY:
This trial is conducted in Asia, Europe and the United States of America (USA). The aim of the trial is to assess the efficacy of concizumab administered s.c. (subcutaneously, under the skin) once daily in preventing bleeding episodes in patients with severe haemophilia A without inhibitors.

ELIGIBILITY:
Inclusion Criteria: - Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine the suitability for the trial - Male patients aged 18 years or older at the time of signing informed consent, diagnosed with severe haemophilia A (FVIII activity below 1%), based on medical records or results at screening Exclusion Criteria: - Known or suspected hypersensitivity to trial product(s) or related products - Known inherited or acquired bleeding disorder other than haemophilia A - Presence of inhibitors (neutralising antibodies) to Factor VIII (equal to or above 0.6 Bethesda Units) at screening measured by the Nijmegen method

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2020-06-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (29):
- United States (5):
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
- France (3):
  - Novo Nordisk Investigational Site, Brest
  - Novo Nordisk Investigational Site, Caen
  - Novo Nordisk Investigational Site, Nantes
- Germany (2):
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Homburg
- Italy (2):
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Rome
- Japan (3):
  - Novo Nordisk Investigational Site, Aichi
  - Novo Nordisk Investigational Site, Nara
  - Novo Nordisk Investigational Site, Tokyo
- Spain (3):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Valencia
- Sweden (2):
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Solna
- Novo Nordisk Investigational Site, Bangkok, Thailand
- Turkey (Türkiye) (4):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, Edirne
  - Novo Nordisk Investigational Site, Istanbul
- Novo Nordisk Investigational Site, Lviv, Ukraine
- United Kingdom (3):
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Derived] Shapiro AD, Angchaisuksiri P, Astermark J, Benson G, Castaman G, Eichler H, Jimenez-Yuste V, Kavakli K, Matsushita T, Poulsen LH, Wheeler AP, Young G, Zupancic-Salek S, Oldenburg J, Chowdary P. Long-term efficacy and safety of subcutaneous concizumab prophylaxis in hemophilia A and hemophilia A/B with inhibitors. Blood Adv. 2022 Jun 14;6(11):3422-3432. doi: 10.1182/bloodadvances.2021006403. PMID 35290453
- [Derived] Shapiro AD, Angchaisuksiri P, Astermark J, Benson G, Castaman G, Chowdary P, Eichler H, Jimenez-Yuste V, Kavakli K, Matsushita T, Poulsen LH, Wheeler AP, Young G, Zupancic-Salek S, Oldenburg J. Subcutaneous concizumab prophylaxis in hemophilia A and hemophilia A/B with inhibitors: phase 2 trial results. Blood. 2019 Nov 28;134(22):1973-1982. doi: 10.1182/blood.2019001542. PMID 31444162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 26 sites in 11 countries as follows: France (3), Germany (2), Italy (1), Japan (3), Spain (3), Sweden (2), Thailand (1), Turkey (3), the United Kingdom (4), Ukraine (1) and the United States (3). In addition to these sites, 5 sites were approved by the IRB/IEC and/or local health authority but did not screen or assign any participants to treatment.
Pre-assignment Details: The trial consisted of two treatment periods: main part which lasted at least 24 weeks for all participants in the trial and an extension part which was up to 102 weeks.
Groups:
- Concizumab: Participants received subcutaneous (s.c.) injection of concizumab once daily for up to 126 weeks (at least 24 weeks main part + 52-102 weeks extension part). The initial dose was 0.15 milligrams per kilogram (mg/kg) and then the dose was escalated to 0.20 and 0.25 mg/kg based on the number of spontaneous bleeding episodes. Participants continued the extension phase at the same dose of concizumab once daily they have reached at the end of main part for 52-102 weeks with the potential dose escalation based on the number of spontaneous bleeding episodes.
Period: Main Period
Arm/Group | Concizumab
Started (Concizumab- Main part) | 36
Full Analysis Set (FAS) | 36
Subject Analysis Set (SAS) | 36
Completed | 32
Not Completed | 4
Not completed — Withdrawal by Subject | 4
Period: Extension Period
Arm/Group | Concizumab
Started | 32
FAS | 32
SAS | 32
Completed | 29
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all dosed participants.
Groups:
- Concizumab: Participants were to receive subcutaneous (s.c.) injection of concizumab once daily for up to 126 weeks (24 weeks main part + 52-102 weeks extension part). The initial dose was 0.15 milligrams per kilogram (mg/kg) and then the dose was escalated to 0.20 and 0.25 mg/kg based on the number of spontaneous bleeding episodes. Participants continued the extension phase at the same dose of concizumab once daily they have reached at the end of main part for 52-102 weeks with the potential dose escalation based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
Arm/Group | Concizumab
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8
  White | 24
  Other | 1
  Not applicable | 3

OUTCOME MEASURES:

1. Primary Outcome: The Number of Bleeding Episodes During at Least 24 Weeks From Treatment Onset
Description: The number of bleeding episodes that were treated during at least 24 weeks from treatment onset are presented. The data is presented while on last dose level when the bleed occurred.
Time Frame: During at least 24 weeks from treatment onset
Population: The FAS included all participants who took al least one dose of the study drug.
Measure: Number; unit: Episodes
Groups:
- Concizumab 0.15 mg/kg- Main Part: Participants received s.c. injection of 0.15 mg/kg concizumab once daily for 24 weeks. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
- Concizumab 0.20 mg/kg- Main Part: Participants received s.c. injection of concizumab once daily for 24 weeks. The initial dose was 0.15 mg/kg which was then escalated to 0.20 mg/kg based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
- Concizumab 0.25 mg/kg- Main Part: Participants received s.c. injection of concizumab once daily for 24 weeks. The initial dose was 0.15 mg/kg which was then escalated to 0.20 and 0.25 mg/kg based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 21 | 7 | 8
Episodes | 43 | 13 | 14

2. Secondary Outcome: The Number of Bleeding Episodes During at Least 76 Weeks From Treatment Onset
Description: The number of bleeding episodes that were treated during at least 76 weeks from treatment onset are presented. The data is presented while on last dose level when the bleed occurred.
Time Frame: During at least 76 weeks from treatment onset
Population: The FAS included all participants who took al least one dose of the study drug.
Measure: Number; unit: Episodes
Groups:
- Concizumab 0.15 mg/kg: Participants were to receive s.c. injection of 0.15 mg/kg of concizumab once daily. Participants who completed the main part (24 weeks) of the study were continued the same dose regimen for concizumab once daily for 52-102 weeks with the potential dose escalation based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
- Concizumab 0.20 mg/kg: Participants were to receive s.c. injection of concizumab once daily. Participants who completed the main part (24 weeks) of the study were continued the same dose regimen for concizumab once daily for 52-102 weeks. The initial dose was 0.15 mg/kg which was then escalated to 0.20 mg/kg based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
- Concizumab 0.25 mg/kg: Participants were to receive s.c. injection of concizumab once daily. Participants who completed the main part (24 weeks) of the study were continued the same dose regimen for concizumab once daily for 52-102 weeks. The initial dose was 0.15 mg/kg which was then escalated to 0.25 mg/kg based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 15 | 10 | 10
Episodes | 67 | 42 | 123

3. Secondary Outcome: The Number of Spontaneous Bleeding Episodes During at Least 24 Weeks From Treatment Onset
Description: Bleeds that were not linked to a specific, known action or event are called spontaneous bleeding episodes. The number of spontaneous bleeding episodes that were treated during at least 24 weeks from treatment onset are presented. The data is presented while on last dose level when the bleed occurred.
Time Frame: During at least 24 weeks from treatment onset
Population: The FAS included all participants who took al least one dose of the study drug.
Measure: Number; unit: Episodes
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 21 | 7 | 8
Episodes | 16 | 8 | 2

4. Secondary Outcome: The Number of Spontaneous Bleeding Episodes During at Least 76 Weeks From Treatment Onset
Description: Bleeds that were not linked to a specific, known action or event are called spontaneous bleeding episodes. The number of spontaneous bleeding episodes that were treated during at least 76 weeks from treatment onset are presented. The data is presented while on last dose level when the bleed occurred.
Time Frame: During at least 76 weeks from treatment onset
Population: The FAS included all participants who took al least one dose of the study drug.
Measure: Number; unit: Episodes
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 15 | 10 | 10
Episodes | 39 | 15 | 29

5. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) During at Least 24 Weeks From Treatment Onset
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product, and which does not necessarily had a causal relationship with this treatment. A TEAE was defined as an event that had onset from the first exposure to treatment until the last visit in the trial. Number of TEAEs that occurred during at least 24 weeks from treatment onset (week 0) are presented. The data is presented per dose level participants were on at the time of onset of the adverse event.
Time Frame: During at least 24 weeks from treatment onset (week 0)
Population: The SAS included all participants who took al least one dose of the study drug.
Measure: Number; unit: Events
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 36 | 15 | 8
Events | 105 | 16 | 9

6. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) During at Least 76 Weeks From Treatment Onset
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product, and which does not necessarily had a causal relationship with this treatment. A TEAE was defined as an event that had onset from the first exposure to treatment until the last visit in the trial. Number of TEAEs that occurred during at least 76 weeks from treatment onset (week 0) are presented. The data is presented per dose level participants were on at the time of onset of the adverse event.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: The SAS included all participants who took al least one dose of the study drug.
Measure: Number; unit: Events
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 36 | 21 | 11
Events | 201 | 53 | 44

7. Secondary Outcome: Occurrence of Anti-concizumab Antibodies During at Least 24 Weeks From Treatment Onset
Description: Occurrence of anti-concizumab antibodies during at least 24 weeks from treatment onset (week 0) is presented. In the reported data, 'Yes' infers number of participants who showed positive anti-concizumab antibody tests whereas 'No' infers number of participants who showed negative anti-concizumab antibody tests.
Time Frame: During at least 24 weeks from treatment onset (week 0)
Population: The FAS included all participants who took al least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Concizumab - Main Part: Participants were to receive subcutaneous (s.c.) injection of concizumab once daily for 24 weeks. The initial dose was 0.15 milligrams per kilogram (mg/kg) and then the dose was escalated to 0.20 and 0.25 mg/kg based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
Arm/Group | Concizumab - Main Part
Number analyzed (Participants) | 36
Participants
  Yes | 3
  No | 33

8. Secondary Outcome: Occurrence of Anti-concizumab Antibodies During at Least 76 Weeks From Treatment Onset
Description: Occurrence of anti-concizumab antibodies during at least 76 weeks from treatment onset (week 0) is presented. In the reported data, 'Yes' infers number of participants who showed positive anti-concizumab antibody tests whereas 'No' infers number of participants who showed negative anti-concizumab antibody tests.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: The FAS included all participants who took al least one dose of the study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Concizumab: Participants who completed main part treatment were continued the same dose regimen for concizumab once daily for 52-102 weeks with the potential dose escalation based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
Arm/Group | Concizumab
Number analyzed (Participants) | 36
Participants
  Yes | 9
  No | 27

9. Secondary Outcome: Change in Fibrinogen During 24 Weeks From Treatment Onset
Description: Change in fibrinogen during 24 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During 24 weeks from treatment onset (week 0)
Population: The SAS included all participants who took al least one dose of the study drug. Overall number of participants analysed = number of participants with available data at the last dose level.
Measure: Mean (Standard Deviation); unit: gram per litre (g/L)
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 19 | 7 | 8
gram per litre (g/L) | -0.08 (0.61) | -0.19 (0.47) | -0.27 (0.29)

10. Secondary Outcome: Change in Fibrinogen During at Least 76 Weeks From Treatment Onset
Description: Change in fibrinogen during at least 76 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: gram per litre (g/L)
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 13 | 10 | 7
gram per litre (g/L) | -0.05 (0.39) | -0.35 (0.56) | -0.23 (0.63)

11. Secondary Outcome: Change in D-dimer During 24 Weeks From Treatment Onset
Description: Change in D-dimer during at least 24 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During 24 weeks from treatment onset (week 0)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 19 | 7 | 8
Nanograms per milliliter (ng/mL) | 184.5 (404.5) | 272.9 (684.4) | 703.8 (693.6)

12. Secondary Outcome: Change in D-dimer During at Least 76 Weeks From Treatment Onset
Description: Change in D-dimer during at least 76 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 14 | 9 | 7
Nanograms per milliliter (ng/mL) | 265.4 (405.3) | 506.7 (369.9) | 1109.3 (818.5)

13. Secondary Outcome: Change in Prothrombin Fragment 1 + 2 (F1 + F2) During 24 Weeks From Treatment Onset
Description: Change in F1 + F2 during 24 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During 24 weeks from treatment onset (week 0)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Picomoles per liter (pmol/L)
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 19 | 7 | 8
Picomoles per liter (pmol/L) | 134 (156) | 257 (524) | 580 (741)

14. Secondary Outcome: Change in Prothrombin Fragment 1 + 2 (F1 + F2) During at Least 76 Weeks From Treatment Onset
Description: Change in F1 + F2 during at least 76 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 14 | 9 | 7
pmol/L | 128 (183) | 211 (207) | 889 (423)

15. Secondary Outcome: Change in Prothrombin Time (PT) During 24 Weeks From Treatment Onset
Description: Change in PT during 24 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During 24 weeks from treatment onset (week 0)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Seconds (sec)
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 19 | 7 | 8
Seconds (sec) | -0.0 (0.4) | -0.3 (0.9) | 0.3 (0.7)

16. Secondary Outcome: Change in Prothrombin Time (PT) During at Least 76 Weeks From Treatment Onset
Description: Change in PT during at least 76 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 14 | 9 | 7
sec | 0.0 (0.4) | 0.8 (2.7) | 0.4 (0.4)

17. Secondary Outcome: Change in Activated Partial Thromboplastin Time (APTT) During 24 Weeks From Treatment Onset
Description: Change in APTT during 24 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During 24 weeks from treatment onset (week 0)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 19 | 7 | 8
sec | 1.5 (10.2) | 3.1 (6.1) | 6.5 (6.9)

18. Secondary Outcome: Change in Activated Partial Thromboplastin Time (APTT) During at Least 76 Weeks From Treatment Onset
Description: Change in APTT during at least 76 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 14 | 9 | 7
sec | 3.1 (4.3) | 9.2 (8.8) | 2.1 (9.4)

19. Secondary Outcome: Change in Anti-thrombin (AT) During 24 Weeks From Treatment Onset
Description: Change in AT during 24 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During 24 weeks from treatment onset (week 0)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Percentage point
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 19 | 7 | 8
Percentage point | 7 (13) | 17 (31) | 7 (18)

20. Secondary Outcome: Change in Anti-thrombin (AT) After at Least 76 Weeks From Treatment
Description: Change in AT after at least 76 weeks from treatment onset (week 0) is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: During at least 76 weeks from treatment onset (week 0)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 14 | 9 | 7
second | 0 (12) | 11 (23) | 15 (25)

21. Secondary Outcome: Concentration of Concizumab Prior to the Last Dose Administration at 24 Weeks
Description: Concentration of concizumab prior to the last dose administration at 24 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration at 24 weeks
Population: The FAS included all participants who took al least one dose of the study drug. Overall number of participants analysed = number of participants with available data at the last dose level.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 18 | 4 | 6
ng/mL | 195.2 (147.0) | 374.4 (644.0) | 2640.8 (4085.6)

22. Secondary Outcome: Concentration of Concizumab Prior to the Last Dose Administration After at Least 76 Weeks
Description: Concentration of concizumab prior to the last dose administration after at least 76 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration after at least 76 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 13 | 10 | 7
ng/mL | 195.1 (161.7) | 392.3 (427.9) | 4015.1 (2902.0)

23. Secondary Outcome: Free Tissue Factor Pathway Inhibitor (TFPI) Concentration Value Prior to the Last Dose Administration at 24 Weeks
Description: Free TFPI (TFPI not bound to concizumab) concentration value prior to the last dose administration at 24 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration at 24 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 18 | 4 | 6
ng/mL | 30.1 (15.6) | 64.4 (35.3) | 12.4 (2.2)

24. Secondary Outcome: Free Tissue Factor Pathway Inhibitor (TFPI) Concentration Value Prior to the Last Dose Administration After at Least 76 Weeks
Description: Free TFPI concentration value prior to the last dose administration after at least 76 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration after at least 76 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 13 | 10 | 7
ng/mL | 26.9 (17.1) | 36.1 (33.1) | 10.1 (5.7)

25. Secondary Outcome: Peak Thrombin Generation Prior to the Last Dose Administration at 24 Weeks
Description: Peak thrombin generation is the maximal concentration of thrombin formed at a given point in time. Peak thrombin generation prior to the last dose administration at 24 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration at 24 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Nanomoles per liter (nmol/L)
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 18 | 4 | 5
Nanomoles per liter (nmol/L) | 88.6 (34.5) | 67.5 (35.0) | 83.4 (10.6)

26. Secondary Outcome: Peak Thrombin Generation Prior to the Last Dose Administration After at Least 76 Weeks
Description: Peak thrombin generation is the maximal concentration of thrombin formed at a given point in time. Peak thrombin generation prior to the last dose administration after at least 76 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration after at least 76 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 13 | 10 | 7
nmol/L | 90.8 (45.2) | 99.1 (36.2) | 111.6 (63.5)

27. Secondary Outcome: Endogenous Thrombin Potential Prior to the Last Dose Administration at 24 Weeks
Description: The endogenous thrombin potential (ETP), defined as the amount of thrombin which can be generated after the in vitro activation of coagulation with tissue factor as trigger and phospholipids as platelet substitute. Endogenous thrombin potential prior to the last dose administration at 24 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration at 24 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Nanomolar*minute (nM*min)
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 18 | 4 | 5
Nanomolar*minute (nM*min) | 1229.1 (340.6) | 965.3 (362.0) | 1176.0 (278.8)

28. Secondary Outcome: Endogenous Thrombin Potential Prior to the Last Dose Administration After at Least 76 Weeks
Description: The endogenous thrombin potential (ETP), defined as the amount of thrombin which can be generated after the in vitro activation of coagulation with tissue factor as trigger and phospholipids as platelet substitute. Endogenous thrombin potential prior to the last dose administration after at least 76 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration after at least 76 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: nM*min
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 13 | 10 | 7
nM*min | 1253.0 (507.3) | 1352.6 (349.5) | 1233.4 (267.9)

29. Secondary Outcome: Thrombin Generation Velocity Index Prior to the Last Dose Administration at 24 Weeks
Description: Thrombin generation velocity index represents the effective rate of thrombin generation between lag time and time to peak. Thrombin generation velocity index prior to the last dose administration at 24 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration at 24 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: nM/min
Arm/Group | Concizumab 0.15 mg/kg- Main Part | Concizumab 0.20 mg/kg- Main Part | Concizumab 0.25 mg/kg- Main Part
Number analyzed (Participants) | 18 | 4 | 5
nM/min | 9.3 (4.8) | 7.0 (5.0) | 8.2 (1.6)

30. Secondary Outcome: Thrombin Generation Velocity Index Prior to the Last Dose Administration After at Least 76 Weeks
Description: Thrombin generation velocity index represents the effective rate of thrombin generation between lag time and time to peak. Thrombin generation velocity index prior to the last dose administration after at least 76 weeks is presented. The data is presented per the last dose level which the participants have reached at the time of assessment.
Time Frame: Prior to the last dose administration after at least 76 weeks
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Nano molar/min (nM/min)
Arm/Group | Concizumab 0.15 mg/kg | Concizumab 0.20 mg/kg | Concizumab 0.25 mg/kg
Number analyzed (Participants) | 13 | 10 | 7
Nano molar/min (nM/min) | 10.3 (6.4) | 10.5 (4.8) | 16.0 (17.1)

ADVERSE EVENTS:
Time Frame: From start of study drug administration (week 0) up to 134 weeks
Description: Results are based on the safety analysis set which included all dosed participants.
  All presented adverse events are treatment emergent adverse events (TEAEs). TEAE was defined as an event that had onset from the first exposure to treatment until the last visit in the trial. The data is presented per dose level participants were on at the time of onset of the adverse event.
  MedDRA version 21.0 is used for the main phase and MedDRA version 22.1 is used for the extension phase.
Groups:
- Concizumab 0.15 mg/kg - Main Part: Participants received s.c. injection of 0.15 mg/kg concizumab once daily for 24 weeks. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
- Concizumab 0.20 mg/kg - Main Part: Participants received s.c. injection of concizumab once daily for 24 weeks. The initial dose was 0.15 mg/kg which was then escalated to 0.20 mg/kg based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
- Concizumab 0.25 mg/kg - Main Part: Participants received s.c. injection of concizumab once daily for 24 weeks. The initial dose was 0.15 mg/kg which was then escalated to 0.20 and 0.25 mg/kg based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
- Concizumab 0.15 mg/kg - Extension Part: Participants were to receive s.c. injection of 0.15 mg/kg of concizumab once daily. Participants who completed the main part (24 weeks) of the study were continued the same dose regimen for concizumab once daily for 52-102 weeks with the potential dose escalation based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
- Concizumab 0.20 mg/kg - Extension Part: Participants were to receive s.c. injection of concizumab once daily. Participants who completed the main part (24 weeks) of the study were continued the same dose regimen for concizumab once daily for 52-102 weeks. The initial dose was 0.15 mg/kg which was then escalated to 0.20 mg/kg based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
- Concizumab 0.25 mg/kg - Extension Part: Participants were to receive s.c. injection of concizumab once daily. Participants who completed the main part (24 weeks) of the study were continued the same dose regimen for concizumab once daily for 52-102 weeks. The initial dose was 0.15 mg/kg which was then escalated to 0.25 mg/kg based on the number of spontaneous bleeding episodes. Breakthrough bleeding episodes occurring to the participants during the trial were treated with turoctocog at home.
Arm/Group | Concizumab 0.15 mg/kg - Main Part | Concizumab 0.20 mg/kg - Main Part | Concizumab 0.25 mg/kg - Main Part | Concizumab 0.15 mg/kg - Extension Part | Concizumab 0.20 mg/kg - Extension Part | Concizumab 0.25 mg/kg - Extension Part
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/15 | 0/8 | 0/19 | 0/14 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/15 | 0/8 | 2/19 | 1/14 | 2/10
Other Adverse Events (participants affected / at risk) | 26/36 | 7/15 | 3/8 | 16/19 | 9/14 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concizumab 0.15 mg/kg - Main Part (N=36) | Concizumab 0.20 mg/kg - Main Part (N=15) | Concizumab 0.25 mg/kg - Main Part (N=8) | Concizumab 0.15 mg/kg - Extension Part (N=19) | Concizumab 0.20 mg/kg - Extension Part (N=14) | Concizumab 0.25 mg/kg - Extension Part (N=10)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concizumab 0.15 mg/kg - Main Part (N=36) | Concizumab 0.20 mg/kg - Main Part (N=15) | Concizumab 0.25 mg/kg - Main Part (N=8) | Concizumab 0.15 mg/kg - Extension Part (N=19) | Concizumab 0.20 mg/kg - Extension Part (N=14) | Concizumab 0.25 mg/kg - Extension Part (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Antithrombin III decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Basophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood fibrinogen decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Crystalluria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 1 (1)
Device physical property issue (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fibrin D dimer increased (Investigations) | 3 (4) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Granuloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemophilic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 7 (7) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 5 (8) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 4 (5) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lip discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 9 (11) | 1 (1) | 0 (0) | 6 (8) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pinguecula (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prothrombin fragment 1.2 increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prothrombin level increased (Investigations) | 3 (4) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyoderma (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soluble fibrin monomer complex increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombin-antithrombin III complex increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tooth repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/97/NCT03196297/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT03196297/SAP_001.pdf